CLINICAL TRIAL: NCT00000635
Title: Treatment of Acyclovir-Resistant Mucocutaneous Herpes Simplex Disease in Patients With AIDS: Open Label Pilot Study of Topical Trifluridine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 172; 11147 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Bacitracin; Polymyxin B; Trifluridine; AIDS-Related Opportunistic Infections; Herpesviridae Infections; Drug Evaluation; Acquired Immunodeficiency Syndrome; Anti-Infective Agents, Local; Antiviral Agents
MeSH Terms: conditions — Herpes Simplex; HIV Infections; AIDS-Related Opportunistic Infections; Herpesviridae Infections; Acquired Immunodeficiency Syndrome | interventions — Trifluridine; bacitracin zinc, neomycin sulfate, polymyxin B, drug combination

INTERVENTIONS:
Drug: Trifluridine
Drug: Bacitracin zinc/Polymyxin B sulfate

SUMMARY:
To determine the safety, effectiveness, and toxicity of topical (local) trifluridine in treating mucocutaneous (at the nasal, oral, vaginal, and anal openings) Herpes simplex virus ( HSV ) disease that has shown resistance to acyclovir in HIV-infected patients. HSV infection in patients with AIDS is often associated with skin sores and frequent recurrences. Treatment with the drug acyclovir results in healing for most patients, but repeated treatment sometimes results in resistance of the virus to acyclovir. Thus, when this happens, other treatments need to be used. Trifluridine is an antiviral drug that is used for the treatment of Herpes infections that occur in the eye. This study attempts to determine if trifluridine is useful for treating HSV sores that have not healed after treatment with acyclovir.

DETAILED DESCRIPTION:
HSV infection in patients with AIDS is often associated with skin sores and frequent recurrences. Treatment with the drug acyclovir results in healing for most patients, but repeated treatment sometimes results in resistance of the virus to acyclovir. Thus, when this happens, other treatments need to be used. Trifluridine is an antiviral drug that is used for the treatment of Herpes infections that occur in the eye. This study attempts to determine if trifluridine is useful for treating HSV sores that have not healed after treatment with acyclovir.

Patients receive at least 10 days (and up to 42 days) of treatment with topical trifluridine. Trifluridine is applied in a thin fluid layer that overlaps the edges of the lesion. Polymyxin B sulfate/bacitracin zinc ointment is then applied over the trifluridine. Lesions are covered by a nonabsorbent dressing. Medication is applied every 8 hours.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Included:

* All medications deemed essential for best patient care, including zidovudine (AZT), Pneumocystis carinii pneumonia (PCP) prophylaxis, and acute or maintenance therapies for other opportunistic infections.

Patients must have the following:

* HIV infection or diagnosis of AIDS.
* Mucocutaneous Herpes simplex virus infection.
* Ability to give informed consent.

Allowed:

* Patients may be co-enrolled in other ACTG studies except for those in which treatments are expected to generate neutropenia. Subjects aged 13 - 17 may be enrolled with appropriate consent from parent or guardian.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Acyclovir, ganciclovir, foscarnet, vidarabine or other investigational drugs with potential anti-Herpes simplex virus activity.

Patients with the following are excluded:

* Previous hypersensitivity reaction to trifluridine, polymyxin B or bacitracin.

Prior Medication:

Excluded:

* Immunomodulators, lymphocyte replacement therapy or biologic response modifiers within 14 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Study Completion 1992-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kessler H A, Study Chair
Locations (8):
- United States (8):
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York

REFERENCES:
- [Background] Kessler H, Weaver D, Benson C, Pottage J, Safrin S, Nevin T, Davis R, Owens S, Korvick J. ACTG 172: treatment of acyclovir-resistant (ACV-R) mucocutaneous herpes simplex virus (HSV) infection in patients with AIDS: open label pilot study of topical trifluridine (TFT). Int Conf AIDS. 1992 Jul 19-24;8(1):We55 (abstract no WeB 1056)
- [Background] Kessler HA, Hurwitz S, Farthing C, Benson CA, Feinberg J, Kuritzkes DR, Bailey TC, Safrin S, Steigbigel RT, Cheeseman SH, McKinley GF, Wettlaufer B, Owens S, Nevin T, Korvick JA. Pilot study of topical trifluridine for the treatment of acyclovir-resistant mucocutaneous herpes simplex disease in patients with AIDS (ACTG 172). AIDS Clinical Trials Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Jun 1;12(2):147-52. doi: 10.1097/00042560-199606010-00007. PMID 8680885